CLINICAL TRIAL: NCT07265661
Title: Surgical Timing After Preoperative Hypofractionated Radiotherapy for Patients With Primary Localized Soft Tissue Sarcoma of the Extremity and Trunk: a Randomized Phase 2 Clinical Trial
Brief Title: Surgical Timing After Preoperative Hypofractionated Radiotherapy for Localized Extremity and Trunk Soft Tissue Sarcoma
Acronym: STARS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STARS
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcoma of the Trunk and Extremities
MeSH Terms: interventions — Aftercare

STUDY DESIGN:
Intervention Model Description: Group A (randomized): hypofractionated radiotherapy (30Gy/5 fractions) and surgical resection at 1-2 weeks after treatment. Group B (randomized): hypofractionated radiotherapy (30Gy/5 fractions) and surgical resection at 4-6 weeks after treatment. Observational cohort: standard treatment with surgery ± standard radiotherapy (50Gy/25 fractions)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): hypofractionated radiotherapy (30Gy/5 fractions) and surgical resection at 1-2 weeks after treatment.
  Interventions: Procedure: hypofractionated radiotherapy (30Gy/5 fractions) and surgical resection at 1-2 weeks after treatment
- Group B (Experimental): hypofractionated radiotherapy (30Gy/5 fractions) and surgical resection at 4-6 weeks after treatment.
  Interventions: Procedure: hypofractionated radiotherapy (30Gy/5 fractions) and surgical resection at 4-6 weeks after treatment
- Observational cohort (No Intervention): Standard treatment with surgery ± standard radiotherapy (50Gy/25 fractions)

INTERVENTIONS:
Procedure: hypofractionated radiotherapy (30Gy/5 fractions) and surgical resection at 1-2 weeks after treatment — hypofractionated radiotherapy (30Gy/5 fractions) and surgical resection at 1-2 weeks after treatment
  Arms: Group A
Procedure: hypofractionated radiotherapy (30Gy/5 fractions) and surgical resection at 4-6 weeks after treatment — hypofractionated radiotherapy (30Gy/5 fractions) and surgical resection at 4-6 weeks after treatment
  Arms: Group B

SUMMARY:
Phase II, national, multicentric, prospective, randomized (1:1) non-inferiority trial with two parallel groups, incorporating a concurrent observational cohort of eligible non-randomized patients, designed to address critical knowledge gaps by prospectively evaluating the safety, efficacy, and feasibility of preoperative ultra-hypofractionated radiotherapy (HFRT) in patients with soft tissue sarcomas (STS) of the extremities and trunk.

DETAILED DESCRIPTION:
This study is designed to address critical knowledge gaps by prospectively evaluating the safety, efficacy, and feasibility of preoperative ultra-hypofractionated radiotherapy (HFRT) in patients with soft tissue sarcomas (STS) of the extremities and trunk. Eligible patients will be randomized to receive an ultra-hypofractionated RT regimen consisting of 30 Gy delivered in 5 fractions of 6 Gy, followed by surgical resection at one of two predefined intervals: either 1-2 weeks or 4-6 weeks after completion of radiotherapy. In parallel, a non-randomized observational cohort will be recorded, consisting of patients treated according to current standard practice - surgery alone or surgery preceded by nonventional RT (50 Gy in 25 fractions) - to provide a contemporaneous benchmark for comparison. The aim of this study is to gather high-quality clinical evidence on the impact of ultra-hypofractionated RT on oncologic outcomes, treatment-related toxicity, perioperative morbidity, and patient-reported quality of life. Evaluation of logistical and economic implications of treatment de-escalation, such as healthcare resource utilization and treatment burden are also an important point to be addressed.

By systematically assessing these endpoints, this study aims to inform future clinical guidelines and support the potential integration of ultra-hypofractionated RT into routine clinical practice for selected patients with localized STS.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent, with the ability to fully understand and effectively communicate, before performance of any study-related procedure not part of normal medical practice, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Age > 18 years
* Proven diagnosis of primary, resectable extremity/trunk wall STS with low-medium risk (Sarculator© predicted 10y-OS > 60%)
* Measurable disease criteria (RECIST 1.1 and CHOI)
* ECOG: 0, 1 or 2 (if influenced by orthopedic condition and not by general status)
* No major contraindication to the planned radiotherapy or surgical treatment
* Active participation with adherence to requested treatment schedule and follow-up
* Female subject will undergo a negative pregnancy test
* Adequate bone marrow function (hemoglobin > 9g/dL, Leukocytes > 3000/mm³, platelets > 100,000/mm³). Patients with plasma creatinine ≤ 1.6 mg/dL, transaminase (AST-SGOT, ALT-SGPT) ≤ 2.5 times the UNL; total bilirubin ≤ 1.5 time the UNL; alkaline phosphatase ≤ 2.5 times the UNL are acceptable. CRP, LDH, total protein and albumin must also be recorded.
* HBV and HCV serologies must be performed prior to patient inclusion. If hepatitis B surface antigen (HBsAg) is positive, further evaluation is required to exclude active viral replication (i.e., testing for hepatitis B e antigen [HBeAg] and HBV DNA). If either of these markers is positive, study inclusion is not recommended. In such cases, prophylactic treatment with lamivudine may be considered at the investigator's discretion. If a potential participant tests positive for anti-HCV antibodies, active infection must be ruled out through a qualitative HCV PCR test. If PCR testing cannot be performed, or if it confirms active infection, the patient will not be eligible for the study. Patients must be HIV-seronegative, with a CD4+ T-cell count greater than 400/mm³. Individuals with clinically significant immunodeficiency-either congenital or acquired-are not eligible for enrollment

Exclusion Criteria:

* Age < 18y
* Soft tissue sarcomas (STS) originating at different sites (i.e., retroperitoneal, abdominal, pelvic, head and neck), gynecological sarcomas, as well as gastrointestinal stromal tumors (GISTs), desmoid-type fibromatosis and pediatric-type sarcomas (i.e., extraosseous Ewing sarcoma, embryonal/alveolar rhabdomyosarcoma, desmoplastic small round cell tumor) are excluded.
* Recurrent or metastatic condition or previous whoop-surgery for sarcoma (incisional biopsies are allowed if performed 6 months before referral).
* Unresectable tumors (with limb sparing surgery)
* Diagnosed oncological condition in the 5 years before enrollment (exceptions: Gleason <6 prostatic adenocarcinoma; In-situ cervical cancer and melanoma; basal cell skin carcinoma radically treated)
* Prior radiation treatment to the site designated for planned surgery or radiotherapy, regardless of indication
* Any medical condition that can impair and reduce life expectancy to less than 2 years including but not limited to significant systemic diseases grade 3 or higher on the CI-CTCAE v5.0 scale, that limit patient availability, or according to investigator judgment may contribute significantly to treatment toxicity
* Uncontrolled bacterial, fungal, or viral infections-either systemic or localized at the site of planned surgery or radiotherapy
* Severe psychiatric disorder, psychological, familial, social or geographic circumstances that limit the patient's ability to comply with the protocol or informed consent.
* Patients who had participated in another clinical trial and/or had received any other investigational product in the last 30 days prior to inclusion
* Patients who had received any other treatment for the disease under study including chemotherapy, radiotherapy, surgery or any other treatment with curative intent. incisional biopsies are allowed if performed 6 months before referral.
* Inability to comply with the requested follow-up
* Women who are pregnant or breast-feeding
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
* BMI > 40 and BMI < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine the incidence of postoperative complications | Day of surgery (DOS); 7-14-21-30-60-90 days post DOS; 4-8-12-16-20-24 months post DOS
  The primary objective of this study is to determine the incidence of postoperative complications (according to Clavien-Dindo) within 90 days from surgery

SECONDARY OUTCOMES:
Quality of Life (QoL) | At last available QoL assessment date for patients without confirmed deterioration
  Quality of Life (QoL)
Overall Survival (OS) | At the last date that patient was known to be alive
  Overall Survival (OS)
Disease-Free Survival (DFS) | Months 4-8-12-16-20-24 post surgery
  Disease-Free Survival (DFS)
Cumulative Incidence of Local Recurrence (CCI-LR) | Months 4-8-12-16-20-24 post surgery
  Cumulative Incidence of Local Recurrence (CCI-LR)
Cumulative Incidence of Distant Metastasis (CCI-DM) | Months 4-8-12-16-20-24 post surgery
  Cumulative Incidence of Distant Metastasis (CCI-DM)
Pathological response | At any time during the study
  Pathological response
Radiological response (RECIST 1.1 and CHOI) | Months 4-8-12-16-20-24 post surgery
  Radiological response (RECIST 1.1 and CHOI)
Treatment-related toxicity | 7-14-21-30-60-90 days DOS, 4-8-12-16-20-24 months post DOS
  Treatment-related toxicity (based on Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 5.0)
Postoperative complications | 7-14-21-30-60-90 days DOS, 4-8-12-16-20-24 months post DOS
  Postoperative complications (classified according to Clavien-Dindo and CCI)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Baia, MD, Principal Investigator — Findazione IRCCS Istituto Nazionale Tumori Milano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cury FL, Viani GA, Gouveia AG, Freire CVS, Grisi GA, Moraes FY. Meta-analysis of 5-day preoperative radiotherapy for soft tissue sarcoma (5D-PREORTS). Radiother Oncol. 2024 Jan;190:109935. doi: 10.1016/j.radonc.2023.109935. Epub 2023 Oct 25. PMID 37884194
- [Background] Guadagnolo BA, Baldini EH. Are We Ready for Life in the Fast Lane? A Critical Review of Preoperative Hypofractionated Radiotherapy for Localized Soft Tissue Sarcoma. Semin Radiat Oncol. 2024 Apr;34(2):180-194. doi: 10.1016/j.semradonc.2023.12.003. PMID 38508783
- [Background] Kosela-Paterczyk H, Teterycz P, Spalek MJ, Borkowska A, Zawadzka A, Wagrodzki M, Szumera-Cieckiewicz A, Morysinski T, Switaj T, Lugowska I, Castaneda-Wysocka P, Zdzienicki M, Goryn T, Rutkowski P. Efficacy and Safety of Hypofractionated Preoperative Radiotherapy for Primary Locally Advanced Soft Tissue Sarcomas of Limbs or Trunk Wall. Cancers (Basel). 2021 Jun 14;13(12):2981. doi: 10.3390/cancers13122981. PMID 34198676
- [Background] Bedi M, Singh R, Charlson JA, Kelly T, Johnstone C, Wooldridge A, Hackbarth DA, Moore N, Neilson JC, King DM. Is 5 the New 25? Long-Term Oncologic Outcomes From a Phase II, Prospective, 5-Fraction Preoperative Radiation Therapy Trial in Patients With Localized Soft Tissue Sarcoma. Adv Radiat Oncol. 2022 Jan 25;7(3):100850. doi: 10.1016/j.adro.2021.100850. eCollection 2022 May-Jun. PMID 35647402
- [Background] Kalbasi A, Kamrava M, Chu FI, Telesca D, Van Dams R, Yang Y, Ruan D, Nelson SD, Dry SM, Hernandez J, Chmielowski B, Singh AS, Bukata SV, Bernthal NM, Steinberg ML, Weidhaas JB, Eilber FC. A Phase II Trial of 5-Day Neoadjuvant Radiotherapy for Patients with High-Risk Primary Soft Tissue Sarcoma. Clin Cancer Res. 2020 Apr 15;26(8):1829-1836. doi: 10.1158/1078-0432.CCR-19-3524. Epub 2020 Feb 13. PMID 32054730
- [Background] Guadagnolo BA, Bassett RL, Mitra D, Farooqi A, Hempel C, Dorber C, Willis T, Wang WL, Ratan R, Somaiah N, Benjamin RS, Torres KE, Hunt KK, Scally CP, Keung EZ, Satcher RL, Bird JE, Lin PP, Moon BS, Lewis VO, Roland CL, Bishop AJ. Hypofractionated, 3-week, preoperative radiotherapy for patients with soft tissue sarcomas (HYPORT-STS): a single-centre, open-label, single-arm, phase 2 trial. Lancet Oncol. 2022 Dec;23(12):1547-1557. doi: 10.1016/S1470-2045(22)00638-6. Epub 2022 Nov 4. PMID 36343656
- [Background] Bishop AJ, Mitra D, Farooqi A, Swanson DM, Hempel C, Willis T, Pearlnath C, Wang WL, Ratan R, Somaiah N, Benjamin RS, Torres KE, Hunt KK, Scally CP, Keung EZ, Satcher RL, Bird JE, Lin PP, Moon BS, Lewis VO, Roland CL, Guadagnolo BA. Moderately hypofractionated, preoperative radiotherapy in patients with soft tissue sarcomas (HYPORT-STS): Updated local control, late toxicities, and patient-reported outcomes. Cancer. 2025 Jan 1;131(1):e35542. doi: 10.1002/cncr.35542. Epub 2024 Aug 27. PMID 39192597
- [Background] Ahmed SK, Xu-Welliver M, Dorr M, Steinert KO, Houdek MT, Rose PS, Karim SM, Ashman JB, Goulding KA, Siontis BL, Haddock MG, Petersen IA. Hypofractionated Preoperative Radiation Therapy for Extremity and Superficial Trunk Soft Tissue Sarcomas: Results of a Prospective, Phase 2 Trial. Int J Radiat Oncol Biol Phys. 2025 Nov 15;123(4):980-989. doi: 10.1016/j.ijrobp.2025.05.006. Epub 2025 May 17. PMID 40389098
- [Background] Kubicek GJ, Kim TW, Gutowski CJ, Kaden M, Eastwick G, Khrizman P, Xu Q, Lackman R. Preoperative Stereotactic Body Radiation Therapy for Soft-Tissue Sarcoma: Results of Phase 2 Study. Adv Radiat Oncol. 2021 Nov 20;7(2):100855. doi: 10.1016/j.adro.2021.100855. eCollection 2022 Mar-Apr. PMID 35387414
- [Background] Rosenberg SA, Tepper J, Glatstein E, Costa J, Baker A, Brennan M, DeMoss EV, Seipp C, Sindelar WF, Sugarbaker P, Wesley R. The treatment of soft-tissue sarcomas of the extremities: prospective randomized evaluations of (1) limb-sparing surgery plus radiation therapy compared with amputation and (2) the role of adjuvant chemotherapy. Ann Surg. 1982 Sep;196(3):305-15. doi: 10.1097/00000658-198209000-00009. PMID 7114936
- [Background] Gronchi A, Miah AB, Dei Tos AP, Abecassis N, Bajpai J, Bauer S, Biagini R, Bielack S, Blay JY, Bolle S, Bonvalot S, Boukovinas I, Bovee JVMG, Boye K, Brennan B, Brodowicz T, Buonadonna A, De Alava E, Del Muro XG, Dufresne A, Eriksson M, Fagioli F, Fedenko A, Ferraresi V, Ferrari A, Frezza AM, Gasperoni S, Gelderblom H, Gouin F, Grignani G, Haas R, Hassan AB, Hecker-Nolting S, Hindi N, Hohenberger P, Joensuu H, Jones RL, Jungels C, Jutte P, Kager L, Kasper B, Kawai A, Kopeckova K, Krakorova DA, Le Cesne A, Le Grange F, Legius E, Leithner A, Lopez-Pousa A, Martin-Broto J, Merimsky O, Messiou C, Mir O, Montemurro M, Morland B, Morosi C, Palmerini E, Pantaleo MA, Piana R, Piperno-Neumann S, Reichardt P, Rutkowski P, Safwat AA, Sangalli C, Sbaraglia M, Scheipl S, Schoffski P, Sleijfer S, Strauss D, Strauss S, Sundby Hall K, Trama A, Unk M, van de Sande MAJ, van der Graaf WTA, van Houdt WJ, Frebourg T, Casali PG, Stacchiotti S; ESMO Guidelines Committee, EURACAN and GENTURIS. Electronic address: clinicalguidelines@esmo.org. Soft tissue and visceral sarcomas: ESMO-EURACAN-GENTURIS Clinical Practice Guidelines for diagnosis, treatment and follow-up☆. Ann Oncol. 2021 Nov;32(11):1348-1365. doi: 10.1016/j.annonc.2021.07.006. Epub 2021 Jul 22. No abstract available. PMID 34303806
- [Background] Callegaro D, Miceli R, Bonvalot S, Ferguson P, Strauss DC, Levy A, Griffin A, Hayes AJ, Stacchiotti S, Pechoux CL, Smith MJ, Fiore M, Dei Tos AP, Smith HG, Mariani L, Wunder JS, Pollock RE, Casali PG, Gronchi A. Development and external validation of two nomograms to predict overall survival and occurrence of distant metastases in adults after surgical resection of localised soft-tissue sarcomas of the extremities: a retrospective analysis. Lancet Oncol. 2016 May;17(5):671-80. doi: 10.1016/S1470-2045(16)00010-3. Epub 2016 Apr 5. PMID 27068860
- [Background] Davis AM, O'Sullivan B, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Hammond A, Benk V, Kandel R, Goddard K, Freeman C, Sadura A, Zee B, Day A, Tu D, Pater J; Canadian Sarcoma Group; NCI Canada Clinical Trial Group Randomized Trial. Late radiation morbidity following randomization to preoperative versus postoperative radiotherapy in extremity soft tissue sarcoma. Radiother Oncol. 2005 Apr;75(1):48-53. doi: 10.1016/j.radonc.2004.12.020. PMID 15948265
- [Background] O'Donnell PW, Griffin AM, Eward WC, Sternheim A, Catton CN, Chung PW, O'Sullivan B, Ferguson PC, Wunder JS. The effect of the setting of a positive surgical margin in soft tissue sarcoma. Cancer. 2014 Sep 15;120(18):2866-75. doi: 10.1002/cncr.28793. Epub 2014 Jun 3. PMID 24894656
- [Background] Haas RL, Floot BGJ, Scholten AN, van der Graaf WTA, van Houdt W, Schrage Y, van de Ven M, Bovee JVMG, van Coevorden F, Vens C. Cellular Radiosensitivity of Soft Tissue Sarcoma. Radiat Res. 2021 Jul 1;196(1):23-30. doi: 10.1667/RADE-20-00226.1. PMID 33914890
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Robba T, Chianca V, Rabino M, Cesaro E, Molea F, Boglione A, Desi GL, Pellegrino P, Boffano M, De Meo S, Merlini A, Santoro F, Linari A, Levis M, Sandrucci S, Comandone A, Grignani G, Piana R, D'Ambrosio L. Sarcopenia is a negative prognostic factor in localized extremities/trunk wall soft tissue sarcomas. Eur J Surg Oncol. 2025 Jul;51(7):109746. doi: 10.1016/j.ejso.2025.109746. Epub 2025 Mar 7. PMID 40120351
- [Background] Fiore M, Ljevar S, Pasquali S, Morelli D, Callegaro D, Sanfilippo R, Barisella M, Sangalli C, Miceli R, Gronchi A. Preoperative Neutrophil-to-Lymphocyte Ratio and a New Inflammatory Biomarkers Prognostic Index for Primary Retroperitoneal Sarcomas: Retrospective Monocentric Study. Clin Cancer Res. 2023 Feb 1;29(3):614-620. doi: 10.1158/1078-0432.CCR-22-2897. PMID 36478176
- [Background] Yoo SK, Fitzgerald CW, Cho BA, Fitzgerald BG, Han C, Koh ES, Pandey A, Sfreddo H, Crowley F, Korostin MR, Debnath N, Leyfman Y, Valero C, Lee M, Vos JL, Lee AS, Zhao K, Lam S, Olumuyide E, Kuo F, Wilson EA, Hamon P, Hennequin C, Saffern M, Vuong L, Hakimi AA, Brown B, Merad M, Gnjatic S, Bhardwaj N, Galsky MD, Schadt EE, Samstein RM, Marron TU, Gonen M, Morris LGT, Chowell D. Prediction of checkpoint inhibitor immunotherapy efficacy for cancer using routine blood tests and clinical data. Nat Med. 2025 Mar;31(3):869-880. doi: 10.1038/s41591-024-03398-5. Epub 2025 Jan 6. PMID 39762425
- [Background] Davis AM, Wright JG, Williams JI, Bombardier C, Griffin A, Bell RS. Development of a measure of physical function for patients with bone and soft tissue sarcoma. Qual Life Res. 1996 Oct;5(5):508-16. doi: 10.1007/BF00540024. PMID 8973131
- [Background] Rossi L, Boffano M, Comandone A, Ferro A, Grignani G, Linari A, Pellegrino P, Piana R, Ratto N, Davis AM. Validation process of Toronto Exremity Salvage Score in Italian: A quality of life measure for patients with extremity bone and soft tissue tumors. J Surg Oncol. 2020 Mar;121(4):630-637. doi: 10.1002/jso.25849. Epub 2020 Jan 19. PMID 31957034